CLINICAL TRIAL: NCT05642442
Title: A 17-week, Phase 2, Randomized, Double-blind, Placebo-controlled, Flexible-dosing, Parallel-group, Multicenter Study of the Efficacy and Safety of Suvecaltamide in the Treatment of Moderate to Severe Residual Tremor in Participants With Parkinson's Disease
Brief Title: A Study of Suvecaltamide in Adults With Moderate to Severe Residual Tremor in Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JZP385-202; 2022-001063-27 (EudraCT Number); 2024-515177-94-00 (EU CTIS Number)
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease; Tremor
Keywords: Suvecaltamide; Moderate tremor; Severe tremor; Parkinson's disease; JZP385; Residual tremor; T-type calcium channels; Movement disorders; Tremor; Parkinson's disease tremor
MeSH Terms: conditions — Parkinson Disease; Tremor; Movement Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants who will receive a matching placebo during the Dose Titration, Optimization Period, and Maintenance Period.
  Interventions: Drug: Placebo
- Sulvecaltamide (Experimental): Participants who will receive an optimal dose of suvecaltamide during the Dose Titration, Optimization Period, and Maintenance Period.
  Interventions: Drug: Suvecaltamide

INTERVENTIONS:
Drug: Placebo — Matching placebo capsule(s) administered every day (QD) orally. Titration may proceed at a rate of 1 matching placebo capsule per day every 7 days as required for optimal efficacy and tolerability up to a maximum number of 3 matching placebo capsules per day.
  Arms: Placebo
Drug: Suvecaltamide — Suvecaltamide capsule administered every day (QD) orally. Titration may proceed at a rate of 10 mg suvecaltamide per day every 7 days as required for optimal efficacy and tolerability up to a maximum dose of 30 mg suvecaltamide per day.
  Other Names: JZP385; CX-8998; MK-8998
  Arms: Sulvecaltamide

SUMMARY:
This is a 17-week double-blind, placebo-controlled, randomized, flexible-dosing, parallel-group, multicenter study designed to evaluate the efficacy and safety of suvecaltamide for the treatment of moderate to severe residual tremor in adult participants with Parkinson's disease (PD). The target population represents participants who have tremor that is not adequately controlled by PD medications and that interferes with their activities of daily living (ADL) and/or with their performance of tasks.

DETAILED DESCRIPTION:
Participants will be randomized 1:1 to receive suvecaltamide or placebo and stratified by the Essential Tremor Rating Scale (TETRAS) composite outcome score (≤ 17 or > 17) as assessed at baseline. The maximum total duration of the study for each participant will be 23 weeks, with a maximum treatment duration of 17 weeks. For each participant, the study consists of a Screening Period (up to 4 weeks), a 5-week Dose Titration and Optimization Period, a 12-week Maintenance Period, and a 2-week Safety Follow-up Period.

ELIGIBILITY:
KEY Inclusion Criteria:

* Diagnosis of clinically probable or clinically established Parkinson's disease (PD) meeting the Movement Disorder Society (MDS) 2015 criteria.
* Participants must be individually optimized on PD medications for the treatment of other cardinal signs of PD (bradykinesia, rigidity) per the judgment of the investigator.
* Participants must be on a stable dosing regimen of their permitted PD and/or other tremor (eg, propranolol) medications for the treatment of motor symptoms for at least 6 weeks prior to screening and do not anticipate the need to make any changes for the duration of the study. A lack of use of medications used to treat motor symptoms also must be stable for 6 weeks prior to screening and remain stable for the duration of the study.
* Participants have moderate to severe impairment associated with tremor at both the screening and baseline visits, as determined by all the following:

  1. A score of > 21 on the TETRAS-ADL subscale; and
  2. CGI-S rating of tremor severity of > 2 (at least moderate for participants ability to function).

KEY Exclusion Criteria:

Medical Conditions

* Female participants who are pregnant, nursing, or lactating or plan to become pregnant during the study or within 90 days of study completion.
* Known history or current evidence of other medical or neurological conditions that may cause or explain the participant's tremor, in the opinion of the investigator, including, but not limited to: psychogenic tremor; myoclonus or ataxia; cerebellar disease; traumatic brain injury; alcohol abuse or withdrawal; mercury poisoning; hyperthyroidism; pheochromocytoma; multiple sclerosis; clinically significant polyneuropathy in the opinion of the investigator; or family history or diagnosis of Fragile X syndrome. Note: Participants with a history of essential tremor are eligible.
* Hoehn & Yahr stage 5 (confinement to bed or wheelchair unless aided).
* Participants who only experience tremor during their "OFF" periods.
* Severity of motor fluctuations or medication-induced dyskinesia that would interfere with the assessment of tremor and/or "ON"/"OFF" periods that are unpredictable per the opinion of the investigator.
* Clinically significant symptomatic orthostatic hypotension in the opinion of the investigator.
* Has evidence at screening of cognitive impairment as defined by a Montreal Cognitive Assessment (MoCA) score < 22 or has a cognitive impairment that, in the investigator's opinion, would prevent completion of study procedures or the ability to provide informed consent.
* History or presence of gastrointestinal disease (including prior bariatric bypass surgery), hepatic (including ALT or AST ≥ 2 × ULN or total bilirubin ≥ 1.5 ULN), or severe renal impairment or end-stage renal disease, or any other condition that, in the opinion of the investigator, may interfere with the absorption, distribution, metabolism, or excretion of suvecaltamide.
* Presence of significant cardiovascular disease at Screening
* History or presence of bipolar and related mood disorders, schizophrenia, schizophrenia spectrum disorders, or other psychotic disorders according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria.

Prior/Concomitant Therapy

* Treatment-naïve patients (ie, those who have never tried PD medication) are excluded from participating in the study.
* Use of PRN medication/substance(s) that might produce or interfere with the evaluation of tremor on study visit days prior to discharge
* Prior or planned surgical intervention to treat PD, including but not limited to magnetic resonance-guided focused ultrasound thalamotomy, deep brain stimulation, ablative thalamotomy, and gamma knife thalamotomy.
* Use of PRN medications to treat tremor or continuous infusion of PD medications. Note: Use of dopaminergic rescue medications (eg, PRN use of carbidopa/levodopa, including levodopa inhalation powder) for non-tremor PD symptoms (eg, rigidity or bradykinesia) is permitted.
* Botulinum toxin injection for the treatment of tremor in the 6 months before screening or planned use at any time during the study. Note: Use of botulinum toxin for other reasons (eg, cosmetic, excessive salivation, dystonia) is permitted as long as the location of use is anatomically distinct from the region with tremor.
* Use of prescription or nonprescription drugs or other products (eg, St. John's Wort) known to be inducers of cytochrome 3A4 (CYP3A4) (cause > 30% reduction of sensitive substrates area under the plasma concentration-time curve [AUC]), which cannot be discontinued at least 4 weeks before baseline, or planned use at any time during the study.
* Use of prescription or nonprescription drugs or other products (eg, grapefruit) known to be strong or moderate inhibitors of CYP3A4, which cannot be discontinued 2 weeks or 5 half-lives, whichever is longer, before baseline, or planned use at any time during the study.
* Use of proton pump inhibitors, which cannot be discontinued at least 2 weeks before baseline, or planned use at any time during the study. (Occasional use of antacids or histamine receptor type 2 [H2] receptor antagonists will be permitted, but antacids should be taken at least 4 hours apart from study intervention; H2 receptor antagonists should be taken at least 4 hours after and/or 12 hours before study intervention).

Diagnostic Assessments

* Known use of recreational drugs, inclusive of the following: phencyclidine, cocaine, opioids, barbiturates, amphetamines, or 3,4-methylenedioxymethamphetamine [ecstasy].
* Opioid use at stable doses, either regularly or PRN, for pain management, as prescribed, is permitted. Use of cannabinoids (including cannabidiol) is permitted if there is no impact on tremor symptoms per the judgment of the investigator.

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jazz Study Director, Study Director — Jazz Pharmaceuticals
Locations (37):
- United States (21):
  - Movement Disorders Center of Arizona, Scottsdale, Arizona
  - Keck School of Medicine of University of Southern California (USC), Los Angeles, California
  - University of Colorado Hospital Anschutz Outpatient Pavilion, Aurora, Colorado
  - Neurology of Central Florida Research Center LLC, Altamonte Springs, Florida
  - Parkinson's Disease and Movement Disorder Center of Boca Raton, Boca Raton, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - USF Parkinson's Disease and Movement Disorders Center, Tampa, Florida
  - NeuroTrials Research Inc., Atlanta, Georgia
  - Hawaii Pacific Health, Honolulu, Hawaii
  - Northwestern Medical Group, Department of Neurology, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, College of Medicine, Department of Neurology, Lexington, Kentucky
  - The Nene and Jamie Koch Comprehensive Movement Disorders Center, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - Dent Neurologic Institute, Amherst, New York
  - Columbia University Irving Medical Center, New York, New York
  - South Shore Neurologic Associates PC, Patchogue, New York
  - University of Cincinnati Gardner Neuroscience Institute (UCGNI), Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Central Texas Neurology Consultants, Round Rock, Texas
  - EverGreenHealth Neuroscience Institute, Kirkland, Washington
- Germany (5):
  - Zentrum f. klinische Forschung Dr. I. Schöll, Bad Homburg
  - Pharmakologisches Studienzentrum Chemnitz GmbH, Chemnitz
  - Curiositas-ad-sanum Beratungs-und Studien GmbH, Haag in Oberbayern
  - Deutsche Klinik fur Diagnostik Helios Klinik Wiesbaden, Hessen
  - Velocity Clinical Research Germany GmbH, Location Wiesbaden, Wiesbaden
- Poland (6):
  - Neurologia Slaska Centrum Medyczne, Katowice
  - Centrum Medyczne Plejady, Krakow
  - Niepubliczny Zaklad Opieki Zdrowotnej Neuromed M.i M. Nastaj Spólka Partnerska, Lublin
  - Maxxmed Centrum Zdrowia i Urody w Lublinie, Lublin
  - Gabinety Lekarskie Rivermed Sp. z o.o., Poznan
  - ETG Neuroscience Sp. z o.o., Warsaw
- Spain (5):
  - Hospital Universitario Cruces, Barakaldo
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: Yes
In accordance with ICMJE requirements, Jazz Pharmaceuticals may provide qualified external researchers access to individual participant data (IPD) and clinical trial data that underlie the results of this trial upon request. Qualified researchers can submit a request on https://www.jazzpharma.com/science/clinical-trial-data-sharing/ as outlined. Jazz Pharmaceuticals reserves the right not to consider a request. For inquiries about Jazz's data sharing policy contact clinicaldatasharing@jazzpharma.com.
URL: https://www.jazzpharma.com/science/clinical-trial-data-sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 169 participants who met all inclusion criteria and no exclusion criteria were enrolled and randomized to treatment at 43 sites in the United States, Germany, Poland, and Spain.
Groups:
- Sulvecaltamide: Participants who received an optimal dose of suvecaltamide during the Dose Titration, Optimization Period, and Maintenance Period.
- Placebo: Participants who received a matching placebo during the Dose Titration, Optimization Period, and Maintenance Period.
Period: Overall Study
Arm/Group | Sulvecaltamide | Placebo
Started | 83 | 86
Completed | 65 | 72
Not Completed | 18 | 14
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 13 | 9
Not completed — Other | 5 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sulvecaltamide | Placebo | Total
Number analyzed (Participants) | 83 | 86 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (7.79) | 67.9 (7.93) | 67.7 (7.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 32 | 54
  Male | 61 | 54 | 115
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 76 | 82 | 158
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 17 on the Essential Tremor Rating Scale (TETRAS) Composite Outcome Score
Description: The TETRAS composite outcome score is the sum of modified items 1 - 11 of the TETRAS-ADL subscale and modified items 6a, 6b, and 7 of the TETRAS-PS. The TETRAS-ADL subscale is a patient-rated scale administered by a trained interviewer that assesses the impact of tremor on day-to-day functioning, such as eating, drinking, dressing, and other fine motor skills. The TETRAS-PS is a clinical rating scale that quantifies tremor in the head, face voice, limbs and trunk. Items 6a, 6b, and 7 of the TETRAS-PS evaluate the impact of upper limb tremor on performance. Each item from the modified subscales ranges from 0 - 3, with 0 representing normal or slightly abnormal and 3 representing severely abnormal. The sum of the 14 items provides the TETRAS composite outcome score, which ranges from 0 - 42, with higher scores representing more severe tremor. The change from baseline is being reported where the greater the change from baseline indicates improvement in outcome.
Time Frame: Baseline to Week 17
Population: Mean TETRAS composite outcome score was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sulvecaltamide | Placebo
Number analyzed (Participants) | 72 | 75
score on a scale | -6.4 (5.39) | -5.3 (5.73)
Statistical Analysis 1: Comparison: Sulvecaltamide vs Placebo; Test type: Superiority; p = 0.2363, Mixed-effect model with repeat measures; Includes baseline TETRAS score, treatment grp, week, treatment grp and baseline by week, randomization strata, and week repeated for each patient; LS mean difference = -1.06, 95% CI 2-sided [-2.83 to 0.70], Standard Error of Mean 0.895

2. Secondary Outcome: Percentage of Participants Who Improved (≥ 1-point Improvement) From Baseline to Week 17 on the Clinical Global Impression of Severity (CGI-S)
Description: The CGI-S is a 5-point Likert-type rating scale assessed by qualified personnel to assess the severity of the impact of tremor in PD on the participants' ability to function. The responses to this investigator-completed scale range from 1 (no limitations) to 5 (severe), with higher scores indicating a worse outcome.
Time Frame: Baseline to Week 17
Population: CGI-S was assessed in participants with available data in the Full Analysis Set.
Measure: Number; unit: percentage of participants
Arm/Group | Sulvecaltamide | Placebo
Number analyzed (Participants) | 72 | 75
percentage of participants | 54.6 | 40.1
Statistical Analysis 1: Comparison: Sulvecaltamide vs Placebo; Test type: Superiority; p = 0.0715, Cochran-Mantel-Haenszel; Adjusted difference (%) = 14.6, 95% CI 2-sided [-1.3 to 30.5] — Adjusted difference of proportions is the weighted average of differences across strata with the CMH weights. Stratification is based on baseline TETRAS Composite Outcome Score

3. Secondary Outcome: Change From Baseline to Week 17 on The Essential Tremor Rating Scale, Activities of Daily Living Subscale (TETRAS-ADL)
Description: The TETRAS-ADL subscale is a patient-rated scale of the impact of tremor on day-to-day functioning administered by a trained interviewer. This subscale directly measures how a patient functions by assessing activities impacted by tremor, such as eating and drinking, dressing and personal hygiene, carrying items, and fine motor skills. The TETRAS-ADL is the sum of 12 items and are rated on a 0 (normal) to 4 (severe) scale. The maximum total score is 48. Higher scores represent more severe tremor. The change from baseline is reported where the greater the change from baseline indicates improvement in outcome.
Time Frame: Baseline to Week 17
Population: TETRAS-ADL was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Sulvecaltamide | Placebo
Number analyzed (Participants) | 72 | 75
score on scale | -7.5 (7.04) | -5.8 (6.48)
Statistical Analysis 1: Comparison: Sulvecaltamide vs Placebo; Test type: Superiority; p = 0.1232, Mixed-effect model with repeat measures; Includes baseline TETRAS-ADL score, treatment grp, week, treatment grp and baseline by week, randomization strata, and week repeated for each patient; LS Mean Difference = -1.68, 95% CI 2-sided [-3.82 to 0.46], Standard Error of Mean 1.084

4. Secondary Outcome: Percentage of Participants Who Improved (≥ 1 Point) From Baseline to Week 17 on the Patient's Global Impression of Severity (PGI-S)
Description: The PGI-S is a 5-point Likert-type rating scale, with response options ranging from 1 (no limitations) to 5 (severe), with higher scores indicating a worse outcome. The participant will rate his/her impression of the severity of the impact of their tremor in PD on their current ability to function.
Time Frame: Baseline to Week 17
Population: PGI-S was assessed in participants with available data in the Full Analysis Set.
Measure: Number; unit: percentage of patients
Arm/Group | Sulvecaltamide | Placebo
Number analyzed (Participants) | 72 | 75
percentage of patients | 54.0 | 43.7
Statistical Analysis 1: Comparison: Sulvecaltamide vs Placebo; Test type: Superiority; p = 0.1906, Cochran-Mantel-Haenszel; Adjusted Difference (%) = 10.5, 95% CI 2-sided [-5.2 to 26.2] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Percentage of Participants Who Were Much Improved on the Patient's Global Impression of Change (PGI-C) at Week 17
Description: The PGI-C is a 5-point Likert-type rating scale that participants use to rate the change in severity of their ability to function due to tremor since baseline. The responses to this scale range from 1 (Much improved) to 5 (Much worse), with higher scores indicating a worse outcome.
Time Frame: Baseline to Week 17
Population: PGI-C was assessed in participants with available data in the Full Analysis Set.
Measure: Number; unit: percentage of patients
Arm/Group | Sulvecaltamide | Placebo
Number analyzed (Participants) | 72 | 75
percentage of patients | 23.9 | 8.2
Statistical Analysis 1: Comparison: Sulvecaltamide vs Placebo; Test type: Superiority; p = 0.0052, Cochran-Mantel-Haenszel; Adjusted difference (%) = 15.6, 95% CI 2-sided [4.7 to 26.6] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Percentage of Participants Who Were Much Improved on the Clinician's Global Impression of Change (CGI-C) at Week 17
Description: The CGI-C is a 5-point Likert-type rating scale that a qualified medical personnel will use to rate the change in severity of the participants' ability to function due to their tremor since baseline. The responses to this scale range from 1 (Much improved) to 5 (Much worse), with higher scores indicating a worse outcome.
Time Frame: Baseline to Week 17
Population: CGI-C was assessed in participants with available data in the Full Analysis Set.
Measure: Number; unit: percentage of patients
Arm/Group | Sulvecaltamide | Placebo
Number analyzed (Participants) | 72 | 75
percentage of patients | 15.7 | 8.1
Statistical Analysis 1: Comparison: Sulvecaltamide vs Placebo; Test type: Superiority; p = 0.1450, Cochran-Mantel-Haenszel; Adjusted Difference (%) = 7.6, 95% CI 2-sided [-2.6 to 17.7] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Change From Baseline to Week 17 on The Essential Tremor Rating Scale, Performance Subscale (TETRAS-PS)
Description: The TETRAS-PS is a clinical rating scale performed by a blinded rater that quantifies tremor in the head, face, voice, limbs, and trunk. Each item will be rated on a scale of 0 (normal) to 4 (severe). The sum of the individual scores provides the overall score, ranging from 0 to 64, with higher scores representing more severe tremor. The change from baseline is being reported with the greater change indicating improvement in outcome.
Time Frame: Baseline to Week 17
Population: TETRAS-PS was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sulvecaltamide | Placebo
Number analyzed (Participants) | 72 | 75
score on a scale | -4.2 (5.41) | -5.9 (6.37)
Statistical Analysis 1: Comparison: Sulvecaltamide vs Placebo; Test type: Superiority; p = 0.1429, Mixed-effect Model With Repeat Measure; Includes baseline TETRAS-PS score, treatment grp, week, treatment grp and baseline by week, randomization strata, and week repeated for each patient; LS Mean Difference = 1.37, 95% CI 2-sided [-0.47 to 3.20]

8. Secondary Outcome: Change From Baseline to Week 17 on TETRAS Total Score (TETRAS-ADL + TETRAS-PS)
Description: The TETRAS total score is the sum of the scores of the full TETRAS-ADL and TETRAS-PS subscales. Each item is rated on a 0 (normal) to 4 (severe) scale, and total scores range from 0 to 112, with higher scores representing more severe tremor. The TETRAS-PS is performed by a blinded rater. The change from baseline is being reported with the greater change indicating an improvement in clinical outcome.
Time Frame: Baseline to Week 17
Population: TETRAS total score was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sulvecaltamide | Placebo
Number analyzed (Participants) | 72 | 75
score on a scale | -11.7 (10.15) | -11.7 (10.48)
Statistical Analysis 1: Comparison: Sulvecaltamide vs Placebo; Test type: Superiority; p = 0.9739, Mixed-effect model with repeat measures; [statistical method as in outcome 1, analysis 1]; Least square mean difference = -0.05, 95% CI 2-sided [-3.35 to 3.24], Standard Error of Mean 1.666

9. Secondary Outcome: Change From Baseline to Week 17 on the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Tremor Score
Description: The MDS-UPDRS tremor score is the sum of selected items from MDS-UPDRS questionnaire Part II (Item 2.10) and 10 items from Part III (Items 3.15a,b, 3.16a,b, 3.17a-e, and 3.18). Item 2.10 assesses the patient report of the presence of tremor and impact on daily activities. Items 3.15, 3.16, and 3.17 are clinician assessments of the amplitude of distinct types of tremor (resting, postural, and kinetic respectively)in the right and left upper extremities separately. Item 3.17 also includes separate clinician assessments for both lower extremities and for the lip/jaw. Item 3.18 provides a clinician assessment of the constancy of rest tremor without regard to anatomical location. The rating for each item ranges from 0 (normal) to 4 (severe) with a maximum possible total MDS-UPDRS tremor score of 44. Higher scores indicate more severe clinical outcome. The change from baseline is being reported with the greater change indicating an improvement in clinical outcome.
Time Frame: Baseline to Week 17
Population: MDS-UPDRS was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sulvecaltamide | Placebo
Number analyzed (Participants) | 65 | 73
score on a scale | -3.5 (3.80) | -3.1 (5.08)
Statistical Analysis 1: Comparison: Sulvecaltamide vs Placebo; Test type: Superiority; p = 0.3029, Mixed-effect model with repeat measures; Includes baseline MDS-UPDR score, treatment grp, week, treatment grp and baseline by week, randomization strata, and week repeated for each patient; Least square mean difference = -0.72, 95% CI 2-sided [-2.09 to 0.65], Standard Error of Mean 0.694

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline up to 14 days after the last dose of study intervention. up to 19 weeks.
Arm/Group | Sulvecaltamide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/86
Serious Adverse Events (participants affected / at risk) | 4/83 | 2/86
Other Adverse Events (participants affected / at risk) | 36/83 | 19/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sulvecaltamide (N=83) | Placebo (N=86)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sulvecaltamide (N=83) | Placebo (N=86)
Urinary tract infection (Infections and infestations) | 3 | 7
Dizziness (Nervous system disorders) | 12 | 7
Somnolence (Nervous system disorders) | 11 | 2
Headache (Nervous system disorders) | 5 | 3
Insomnia (Psychiatric disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT05642442/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT05642442/SAP_001.pdf